CLINICAL TRIAL: NCT00000853
Title: A Phase I, Multicenter, Randomized, Double-Blind, Placebo-Controlled HIV-1 Vaccine Trial to Evaluate the Safety and Immunogenicity of Low Dose MN rsgp120/HIV-1 (Genentech) in Combination With QS21 Adjuvant or Alum in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 016B; 10566 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: rgp120/HIV-1MN

SUMMARY:
To expand the safety information regarding MN rsgp 120/HIV-1 formulated with QS21 or alum. To evaluate the immunogenicity of low doses of MN rsgp 120/HIV-1 formulated with QS21 or alum.

Studies to date indicate that there may be a dose-sparing effect with the use of QS21. In animal studies, when QS21 has been employed as an adjuvant, it shifted both the dose response curve and allowed less antigen to elicit equivalent binding antibody titers to the rgp120 protein. There may also be an acceleration in the course of antibody response after both the first and the second immunizations. Although the final titers in response to vaccine given in both alum and QS21 appear similar after 3 doses in humans, this plateau may be reached more readily, and with a lower antigen dose, when using QS21 as an adjuvant. In addition, it has been established that using a lower dose of antigen may elicit an immune response which is characterized by lymphoproliferation and production of TH1-like cytokines such as INF-gamma, interleukin-2, interleukin-4, interleukin-5 and interleukin-10.

DETAILED DESCRIPTION:
Studies to date indicate that there may be a dose-sparing effect with the use of QS21. In animal studies, when QS21 has been employed as an adjuvant, it shifted both the dose response curve and allowed less antigen to elicit equivalent binding antibody titers to the rgp120 protein. There may also be an acceleration in the course of antibody response after both the first and the second immunizations. Although the final titers in response to vaccine given in both alum and QS21 appear similar after 3 doses in humans, this plateau may be reached more readily, and with a lower antigen dose, when using QS21 as an adjuvant. In addition, it has been established that using a lower dose of antigen may elicit an immune response which is characterized by lymphoproliferation and production of TH1-like cytokines such as INF-gamma, interleukin-2, interleukin-4, interleukin-5 and interleukin-10.

Patients will be recruited and screened and those determined as eligible will be enrolled in the study. Initially, 5 patients will be randomized into each combination of MN rsgp 120/HIV-1 dose and adjuvant, QS21 or alum, along with 2 controls for each adjuvant group. An additional 10 patients will be randomized equally between the QS21 and alum arms to the lowest dose group having 2 or more responders defined as an MN Vital Dye neutralization titer greater than or equal to 10 measured at 2 weeks after the second vaccination. 1 additional control will also be randomized to each adjuvant group. If neither dose has 2 or more responders, no additional patients will be enrolled. Patients will receive their randomly assigned injections at months 0, 1 and 6. Patients will be tested for DTH to MN rsgp 120 at 12 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have or be:

* Healthy.
* Negative ELISA for HIV.
* Negative for Hepatitis B surface antigen.
* Normal urine dipstick.
* Normal history and physical examination.
* Availability for 18 months of follow-up.

Risk Behavior: Required:

* Lower-risk sexual behavior as defined by AVEG.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Medical or psychiatric condition or occupational responsibilities, which preclude subject compliance with the protocol (e.g., recent suicidal ideation or present psychosis).
* Active syphilis. NOTE: If the serology is documented to be false positive due to a remote (> 6 months) treated infection, the volunteer is eligible).
* Active tuberculosis. NOTE: Volunteers with a positive PPD and a normal chest X-ray showing no evidence of TB and not requiring INH therapy are eligible.

Patients with any of the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, malignancy, autoimmune disease.
* History of cancer unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of cure.
* History of anaphylaxis or history of other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care.
* History of suicide attempts or past psychosis.
* History of reaction to thimerosal.

Prior Medication:

Excluded:

* History of use of immunosuppressive medication.
* Live attenuated vaccines within 60 days of study. NOTE: Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 2 weeks away from HIV immunizations.
* Use of experimental agents within 30 days prior to study.
* Prior receipt of HIV-1 vaccines or placebo recipient in previous HIV vaccine trial.

Prior Treatment:

Excluded:

* Receipt of blood products or immunoglobulin in the past 6 months.

Risk Behavior:

Excluded:

* Subjects with identifiable higher-risk behavior for HIV infection as determined by screening questionnaire designed to identify risk factors for HIV infection.
* History of injection drug use within the last 12 months prior to enrollment.
* Higher- or intermediate-risk sexual behavior as defined by AVEG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Study Completion 1999-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McElrath J, Study Chair; Evans T, Study Chair
Locations (3):
- United States (3):
  - UAB AVEG, Birmingham, Alabama
  - Univ. of Rochester AVEG, Rochester, New York
  - UW - Seattle AVEG, Seattle, Washington

REFERENCES:
- [Background] Zolla-Pazner S, Alving C, Belshe R, Berman P, Burda S, Chigurupati P, Clements ML, Duliege AM, Excler JL, Hioe C, Kahn J, McElrath MJ, Sharpe S, Sinangil F, Steimer K, Walker MC, Wassef N, Xu S. Neutralization of a clade B primary isolate by sera from human immunodeficiency virus-uninfected recipients of candidate AIDS vaccines. J Infect Dis. 1997 Apr;175(4):764-74. doi: 10.1086/513969. PMID 9086128